CLINICAL TRIAL: NCT00449306
Title: Physical,Histological,and Genetic Analyses of Lipid-rich Atherosclerotic Plaques
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: University Hospital Goettingen (Other); Carmel Medical Center (Other); CVPath Institute Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: SHEBA-01-2354-JS-CTIL
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Atherosclerosis; Aortic Aneurysm; Peripheral Vascular Diseases
Keywords: Atherosclerosis; Carotid plaque; Abdominal aortic aneurysm; Vulnerable plaque; Angiogenesis; Intraplaque hemorrhage; Carotid artery atherosclerosis
MeSH Terms: conditions — Atherosclerosis; Aortic Aneurysm; Peripheral Vascular Diseases; Aortic Aneurysm, Abdominal; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Tissue for RNA extraction (frozen); Tissue for histological analysis (formalin fixation); Plasma for CV biomarkers (frozen)
Oversight: Data Monitoring Committee: No

SUMMARY:
Lipid-rich atherosclerotic plaques, or "vulnerable plaques" are prone to rupture, causing local intravascular thrombosis, with subsequent grave clinical consequences. Atherosclerotic plaques normally removed during surgery, and peripheral blood samples will be studied to achieve the following objectives:

"1" Define histological features of the vulnerable plaque, analyze its physical characteristics, and investigate selected gene expression.

"2" Study biomarkers of inflammation in conjunction with the presence of vulnerable plaques.

"3" Explore the potential role of infection in atherogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of symptomatic carotid stenosis exceeding 60%(TIAs or stroke within the last 6 months), and asymptomatic carotid artery stenosis (presenting with progressive carotid stenosis, exceeding 70%)
* Abdominal aortic aneurysm, and aortic occlusive disease
* Peripheral occlusive or aneurysmal disease

Exclusion Criteria:

* Non-compliant patients, incapable of granting approval by informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic patients
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2001-03; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
To uncover mechanisms of cardiovascular diseases | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Schneiderman, MD, Principal Investigator — Department of Vascular Surgery, Sheba Medical Center, Tel Hashomer
Locations (1):
- Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel

REFERENCES:
- [Derived] Ben-Zvi D, Savion N, Kolodgie F, Simon A, Fisch S, Schafer K, Bachner-Hinenzon N, Cao X, Gertler A, Solomon G, Kachel E, Raanani E, Lavee J, Kotev Emeth S, Virmani R, Schoen FJ, Schneiderman J. Local Application of Leptin Antagonist Attenuates Angiotensin II-Induced Ascending Aortic Aneurysm and Cardiac Remodeling. J Am Heart Assoc. 2016 May 3;5(5):e003474. doi: 10.1161/JAHA.116.003474. PMID 27143353
- [Derived] Schneiderman J, Schaefer K, Kolodgie FD, Savion N, Kotev-Emeth S, Dardik R, Simon AJ, Halak M, Pariente C, Engelberg I, Konstantinides S, Virmani R. Leptin locally synthesized in carotid atherosclerotic plaques could be associated with lesion instability and cerebral emboli. J Am Heart Assoc. 2012 Oct;1(5):e001727. doi: 10.1161/JAHA.112.001727. Epub 2012 Oct 25. PMID 23316287